CLINICAL TRIAL: NCT02696616
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses of BI 655088 Administered by Intravenous Infusion in Healthy Male Subjects (Single-blind, Partially Randomised Within Dose Groups, Placebo-controlled, Parallel Group Design)
Brief Title: Single Rising Dose Study of BI 655088 Administered Intravenously in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1339.1; 2014-002413-29 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- BI 655088 (Experimental)
  Interventions: Drug: BI 655088
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 655088
  Arms: BI 655088
Drug: Placebo
  Arms: Placebo

SUMMARY:
Investigation of safety and tolerability of BI 655088 following intravenous infusion of single rising doses and exploration of the pharmacokinetics and pharmacodynamics of BI 655088 after single dosing

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects
* Age of 18 to 50 years
* Body mass index (BMI) of 18.5 to 29.9 kg/m2
* Additional inclusion criteria may apply

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg or diastolic blood pressure outside the range of 50 to 90 mmHg or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures and stroke), and other relevant neurological disorders or psychiatric disorders
* Additional exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-rising dose trial, partially randomised within dose groups, placebo-controlled, single-blind, parallel-group design with 6 dose groups.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that the subjects met all strictly implemented inclusion and none of the exclusion criteria. Subjects would not have been treated with the trial treatment if any one of the specific entry criteria had been violated.
Groups:
- Placebo: Comparator product: Matching Placebo to BI 655088 (buffer solution).
  Mode of administration: Intravenous (IV) infusion for 120 minutes
- BI 655088 2 mg: BI investigational product: Single Dose of 2 milligram (mg) of BI 655088 as solution for infusion (10 mg/millilitre (mL) in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- BI 655088 6 mg: BI investigational product: Single Dose of 6mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- BI 655088 20 mg: BI investigational product: Single Dose of 20mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- BI 655088 50 mg: BI investigational product: Single Dose of 50mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- BI 655088 100 mg: BI investigational product: Single Dose of 100mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- BI 655088 200 mg: BI investigational product: Single Dose of 200mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
Period: Overall Study
Arm/Group | Placebo | BI 655088 2 mg | BI 655088 6 mg | BI 655088 20 mg | BI 655088 50 mg | BI 655088 100 mg | BI 655088 200 mg
Started | 12 | 5 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 4 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set:
  This subject set included all subjects who were documented to have received at least
  1 dose of trial drug. It was used for analysis of safety, demographic data, and baseline characteristics, and disposition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 655088 2 mg | BI 655088 6 mg | BI 655088 20 mg | BI 655088 50 mg | BI 655088 100 mg | BI 655088 200 mg | Total
Number analyzed (Participants) | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (8.5) | 42.0 (9.4) | 33.0 (5.0) | 42.3 (7.5) | 43.7 (6.3) | 34.0 (9.7) | 37.8 (9.5) | 38.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 5 | 6 | 6 | 6 | 6 | 6 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 10 | 4 | 6 | 6 | 5 | 6 | 5 | 42
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events
Description: The number of subjects with drug-related adverse events.
Time Frame: up to 99 days after start of drug administration
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Placebo | BI 655088 2 mg | BI 655088 6 mg | BI 655088 20 mg | BI 655088 50 mg | BI 655088 100 mg | BI 655088 200 mg
Number analyzed (Participants) | 12 | 5 | 6 | 6 | 6 | 6 | 6
Participants | 2 | 1 | 2 | 1 | 0 | 0 | 0

2. Secondary Outcome: Maximum Measured Concentration of BI 655088 in Plasma (Cmax)
Description: Maximum measured concentration of BI 655088 in plasma (Cmax).
  Time frame for all dose groups: within 3 hours before and 10, 24, 36, 48, 72, 96, 120, 144, 168, 264, 336, 432, 504, 600, 672, 840, 1008, 1176, 1344, 1512, 1680 and 2016 hours following start of infusion. In additional, the following time points for the 2 milligram group: 0.25, 0.5, 1, 1.5, 2.25, 2.5, 3, 6, 8, 12 and 30 hours following start of infusion.
Time Frame: Up to 2016 hours. See endpoint description for a detailed timeframe.
Population: Pharmacokinetic (PK) parameter analysis set:
  This subject set included all subjects who were documented to have received at least
  1 dose of BI 655088 and who provided at least 1 PK endpoint value that was not excluded (due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg) / millilitre (mL)
Arm/Group | BI 655088 2 mg | BI 655088 6 mg | BI 655088 20 mg | BI 655088 50 mg | BI 655088 100 mg | BI 655088 200 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
microgram (µg) / millilitre (mL) | 0.593 (8.98) | 1.69 (15.8) | 5.76 (24.9) | 13.1 (12.5) | 17.3 (66.2) | 48.8 (4.90)

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 655088 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz (area under the concentration-time curve of BI 655088 in plasma over the time interval from 0 to the last quantifiable data point).
  Time frame for all dose groups: within 3 hours before and 10, 24, 36, 48, 72, 96, 120, 144, 168, 264, 336, 432, 504, 600, 672, 840, 1008, 1176, 1344, 1512, 1680 and 2016 hours following start of infusion. In additional, the following time points for the 2 milligram group: 0.25, 0.5, 1, 1.5, 2.25, 2.5, 3, 6, 8, 12 and 30 hours following start of infusion.
Time Frame: Up to 2016 hours. See endpoint description for a detailed timeframe.
Population: Pharmacokinetic (PK) parameter analysis set: This subject set included all subjects who were documented to have received at least 1 dose of BI 655088 and who provided at least 1 PK endpoint value that was not excluded (due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability). 1 subject was excluded from the 200 mg group due to missing samples after 840 hours.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg)∙hour (h)/millilitre (mL)
Arm/Group | BI 655088 2 mg | BI 655088 6 mg | BI 655088 20 mg | BI 655088 50 mg | BI 655088 100 mg | BI 655088 200 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5
microgram (µg)∙hour (h)/millilitre (mL) | 12.5 (22.8) | 63.8 (13.2) | 392 (21.2) | 1250 (17.0) | 2360 (124) | 7210 (18.3)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 655088 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: AUC0-∞ (area under the concentration-time curve of BI 655088 in plasma over the time interval from 0 extrapolated to infinity).
  Time frame for all dose groups: within 3 hours before and 10, 24, 36, 48, 72, 96, 120, 144, 168, 264, 336, 432, 504, 600, 672, 840, 1008, 1176, 1344, 1512, 1680 and 2016 hours following start of infusion. In additional, the following time points for the 2 milligram group: 0.25, 0.5, 1, 1.5, 2.25, 2.5, 3, 6, 8, 12 and 30 hours following start of infusion.
Time Frame: Up to 2016 hours. See endpoint description for a detailed timeframe.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg)∙hour (h) /millilitre(mL)
Arm/Group | BI 655088 2 mg | BI 655088 6 mg | BI 655088 20 mg | BI 655088 50 mg | BI 655088 100 mg | BI 655088 200 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
microgram (µg)∙hour (h) /millilitre(mL) | 12.9 (24.4) | 65.7 (11.9) | 395 (21.3) | 1250 (17.0) | 2360 (124) | 7010 (17.9)

ADVERSE EVENTS:
Time Frame: from individual subjects' drug administration until individual subjects' end of trial ,up to 99 days
Description: Treated set: This subject set included all subjects who were documented to have received at least 1 dose of trial drug.
Groups:
- 2 mg BI: BI investigational product: Single Dose of 2 milligram (mg) of BI 655088 as solution for infusion (10 mg/millilitre (mL) in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- 6 mg BI: BI investigational product: Single Dose of 6mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- 20 mg BI: BI investigational product: Single Dose of 20mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- 50 mg BI: BI investigational product: Single Dose of 50mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- 100 mg BI: BI investigational product: Single Dose of 100mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
- 200 mg BI: BI investigational product: Single Dose of 200mg of BI 655088 as solution for infusion (10 mg/mL in buffer solution).
  Mode of administration: IV infusion for 120 minutes
Arm/Group | Placebo | 2 mg BI | 6 mg BI | 20 mg BI | 50 mg BI | 100 mg BI | 200 mg BI
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/5 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 10/12 | 4/5 | 3/6 | 2/6 | 1/6 | 2/6 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | 2 mg BI (N=5) | 6 mg BI (N=6) | 20 mg BI (N=6) | 50 mg BI (N=6) | 100 mg BI (N=6) | 200 mg BI (N=6)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pathogen resistance (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | 2 mg BI (N=5) | 6 mg BI (N=6) | 20 mg BI (N=6) | 50 mg BI (N=6) | 100 mg BI (N=6) | 200 mg BI (N=6)
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT02696616/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT02696616/SAP_001.pdf